CLINICAL TRIAL: NCT04357561
Title: Investigation of The Effects of Scoliosis Specific Exercises Before Adolescent Idiopathic Scoliosis Surgery
Brief Title: The Effects of Scoliosis-Specific Exercises Before Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Tugce Ozen, Research Assistant, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 092019939
Record Dates: First submitted 2020-04-15; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; preoperative rehabilitation; surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Schroth best practice) (Experimental): Exercise program will consists of scoliosis-specific exercises (schroth best practice), which is a pattern specific scoliosis rehabilitation concept and provide three dimensional improvements and include patient education for maintaining corrected posture in daily life. In addition, these exercises provide improvements in neuromuscular control and the endurance of the postural muscles.
  Interventions: Behavioral: Exercise group (Schroth best practice)
- Control group (No Intervention): Due to there is not a standard preoperative exercise protocol, additional exercise program will not be applied in control group. The patients will wait for the surgery in their routine daily life. Measurements will be performed at the same time frame in experimental group.

INTERVENTIONS:
Behavioral: Exercise group (Schroth best practice) — Exercise program will be structured with scoliosis specific exercises (schroth best practice). Schroth best pratice is a pattern spesific scoliosis rehabilitation concept which aimes active self correction during curve pattern specific curve activities of daily life. Exercises for rotational breathing, everyday activities, spinal mobilization and corrective exercises will be specified based on the curve type and applied under the supervision of a physiotherapist.
  Arms: Exercise group (Schroth best practice)

SUMMARY:
The aim of this study is to investigate the effects of scoliosis-specific exercises in adolescent idiopathic scoliosis patients, who had surgical indication, on functional capacity, cosmetic deformity perception, quality of life in postoperative period.

DETAILED DESCRIPTION:
30 adolescent idiopathic scoliosis patients, who had surgery indication and aged between 10-18 years, will be included. The participants will be randomised into two groups. 15 patients will be included in the exercise group and 15 patients in the control group. In the exercise group, a total of 12 sessions of exercise are planned, 6 weeks before the surgery and 2 days per week. In the control group, the exercise protocol will not be performed before surgery.

The outcomes will include the cosmetic deformity, quality of life, pain level, functional capacity, spine flexibility. In the exercise group, the evaluations will be made in the first interview (before exercise application), at the end of 6 weeks of exercise (when the exercise program is completed), in the early postoperative period and 12 weeks after surgery. Evaluations in the control group will be carried out at the first interview, at the 6th week, in the early postoperative period, and at the 12th week postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with adolescent idiopathic scoliosis
* Aged between 10 and 18 years
* To have surgery indication

Exclusion Criteria:

* Leg discrepancy
* Cervical region participation to curve
* Additional disease may cause respiratory problem

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Functional performance | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Six-minute walking test will be used. The patients will be asked to walk at his/her own pace of walking in a 30 meter course. The distance walked over a span of 6 minutes will be recorded.
Pain perception | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Pain level will be evaluated with visual analog scale. Patients will be asked to indicate their pain level in activity and in rest period.
Health related quality of life | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Scoliosis Research Society-30 will be used for quality of life evaluation. This questionnaire consists of 30 questions, scored between 1 and 5, and evaluate pain, function, self-image, mental health and treatment satisfaction.
  Pediatric Quality of Life Inventory is a self-report questionnaire developed for children and their families. consists of 22 questions and evaluate physical and psychosocial health. Higher scores indicate better quality of life.
Cosmetic deformity perception | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Walter Reed Visual Assessment Scale-Walter Reed Visual Assessment Scale will be used to evaluate individuals' self-perception of cosmetic deformities and the effectiveness of treatment in improving body cosmetic deformity. It focuses on the person's perception of posture and the severity of the curve. This questionnaire is divided into 7 parameters including body curvature, rib prominence, waist prominence, head-rib-pelvis positional relation, head-pelvis relation, shoulder level and scapula rotation. Each parameter is scored from 1 to 5.
Spine flexibility | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Forward bending test will be applied. The patient is asked to reach the feet with his hands while sitting on a hard floor with both feet extended, with feet 15 cm apart from each other, based on a 25 cm long step, without bringing the knees flexed. measured and saved as centimeter.
  Side bending test will be used to measure the flexibility of spine in right and left lateral flexion. The patient is asked to bend his back to the right and left sides, without separating his back from the wall. The result sill be recorded as centimeter.
Trunk rotation | Change from baseline at week 6, postoperative 4.week, postoperative 12.week
  Trunk rotation will be measured with scoliometer while the patient is in forward bending position with barefoot. The highest value in each part will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tugce Ozen, MSc, Principal Investigator — Research Assistant
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No